CLINICAL TRIAL: NCT03910257
Title: the Effectiveness of Nutrition Education Module to Knowledge of Preschooler Children in Public Kindergarten at 3 Districts of Riau Province
Brief Title: Nutrition Education Module for Preschooler Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Responsible Party: Principal Investigator, Muharni Harahap, Affiliated Researcher, SEAMEO Regional Centre for Food and Nutrition
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: modul gizi
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Children Who Registered on the Selected Public Kindergarten and Agree to Follow the Study Assigned by Their Parents and Teacher

STUDY DESIGN:
Intervention Model Description: a quasi-experimental research design with pre-and post-test control group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nutrition education module (Experimental): 12 activities of the nutrition education module pre and post test
  Interventions: Behavioral: nutrition education module
- control group (No Intervention): no intervention pre and post test

INTERVENTIONS:
Behavioral: nutrition education module — 12 activities of nutrition education module will deliver by the teacher. The activities consists of coloring my meal plate, playing pictures, story telling: Zizi and Ziko, pictures station, fruits and vegetables card, cooking class, planting bean sprouts, field visit to fruits and vegetables garden, making collages, dot to dot, watching video, making healthy snacks
  Arms: nutrition education module

SUMMARY:
This study evaluates the knowledge of preschooler children before and after intervention of nutrition education using nutrition education module for preschooler children. The teachers will be given training regarding the module and deliver it in the class during the intervention.

DETAILED DESCRIPTION:
A nutrition education module for preschooler children had been developed in the previous study. The module consists of 3 topics of nutrition (my meal plate, fruits and vegetables, healthy snacks). Each topic consists of 4 activities engaging children and teachers. A total of 12 activities will be delivered on 4 consecutive school day every week.

The teacher will deliver the nutrition education which trained prior to the study.

ELIGIBILITY:
Inclusion Criteria:

* children registered in selected public kindergarten
* grade/class B kindergarten
* willing to follow the study

Exclusion Criteria:

-

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Changes on nutrition related knowledge before and after intevention | 3 weeks
  a self administered structured questionnaire regarding nutrition related knowledge (my meal plate, fruits and vegetables, healthy snacks) using pictures yielding a total score between 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- TK Negeri Pembina Pekanbaru, Pekanbaru, Riau, Indonesia

IPD SHARING:
Plan to Share IPD: Yes